CLINICAL TRIAL: NCT05896215
Title: A Phase II Clinical Study of KNP2002 Ointment in Patients With Common Warts (OM202JA)
Brief Title: OM202JP Clinical Study of KNP2002
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KinoPharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OM202JA
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-04

CONDITIONS: Common Wart
Keywords: Common Wart
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Low dose group (Experimental): Topical administration of low dose of KPN2002
  Interventions: Drug: KNP2002
- Middle dose group (Experimental): Topical administration of middle dose of KPN2002
  Interventions: Drug: KNP2002
- High dose group (Experimental): Topical administration of high dose of KPN2002
  Interventions: Drug: KNP2002
- Placebo group (Placebo Comparator): Topical administration of placebo
  Interventions: Drug: Placebo of KNP2002

INTERVENTIONS:
Drug: KNP2002 — Dairy topical administration for 12 weeks
  Other Names: KV-0132
  Arms: High dose group; Low dose group; Middle dose group
Drug: Placebo of KNP2002 — Dairy topical administration for 12 weeks
  Arms: Placebo group

SUMMARY:
The goal of this clinical trial is to evaluate safety and efficacy of KNP2002 in patients with common warts aged 15 to 50 years old.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 15 to 49 years old
* Subjects with common warts on the upper or lower limb
* Subjects who agree to contraception from obtaining consent to 4 weeks after the end of administration
* Subjects who have given their voluntary written consent to participate in this clinical trial

Exclusion Criteria:

* Subjects with 5 or more warts on the upper or lower limbs
* Subjects who are scheduled to undergo treatment such as physical therapy or chemotherapy for warts
* Subjects with a history of allergy to topical skin preparations
* Subjects with a history of malignant tumor within 5 years before administration of study drug
* Subjects with any of the following diseases: Malignant tumor; Serious heart disease; Poorly controlled diabetes/hypertension
* Women who are pregnant, may become pregnant, or are breastfeeding

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 159 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2024-07-27 (Actual); Study Completion 2024-07-27 (Actual)

PRIMARY OUTCOMES:
Change in wart area | At 16 weeks after starting administration
  Percent change in wart area from baseline

SECONDARY OUTCOMES:
Change in wart area over time | At 4, 8, 12, and 16 weeks after starting administration
  Percent change in wart area from baseline
Wart improvement rate | At 4, 8, 12, and 16 weeks after starting administration
  Wart improvement rate categorized by rate of change in wart area
Wart disappearance rate | Up to 16 weeks after starting administration
  Proportion of patients with warts disappearing

CONTACTS AND LOCATIONS:
Locations (15):
- Japan (15):
  - Kawaharamachi Dermatology, Maebashi, Gunma
  - Tetsuya Dermatology, Himeji, Hyōgo
  - Takashima Dermatology, Kobe, Hyōgo
  - Nishino Dermatology Clinic, Kobe, Hyōgo
  - Queen's Square, Dermatology, Allergy, Yokohama, Kanagawa
  - Asai Dermatology Clinic, Yokohama, Kanagawa
  - Okawa Dermatology Clinic, Sakai, Osaka
  - Sugai Dermatology Parkside Clinic, Utsunomiya, Tochigi
  - Tsunoda Clinic, Arakawa-Ku, Tokyo
  - Sugisawa Dermatology Clinic, Katsushika-ku, Tokyo
  - Igarashi Clinic, Kita-ku, Tokyo
  - Maruyama Dermatology Clinic, Koto-Ku, Tokyo
  - Todoroki Dermatology Clinic, Nakano-Ku, Tokyo
  - Okuda Dermatology Clinic, Setagaya-Ku, Tokyo
  - Hayami Dermatology, Osaka

IPD SHARING:
Plan to Share IPD: No